CLINICAL TRIAL: NCT07237282
Title: A Phase 1 Clinical Trial of Adjuvanted Protein-based HCV Vaccine Candidates (HCV Vaccine Trial)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00147152
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hepatitis C
Keywords: Vaccine
MeSH Terms: conditions — Hepatitis C | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: The trial is divided into 2 stages - the 1st stage will be an open-label sentinel safety dosing in 3 participants; if no significant attributable safety concerns after these first 3 participants have received doses 1 and 2 and had their followup; the 2nd stage will be a double-blinded, placebo-controlled, randomized control trial with AVIHepC1 (the newly formulated E1E2 vaccine) compared to saline control in 24 volunteers (12 per trial arm) for a total of 27 participants.
  Participants will receive doses of the investigational product (AVIHepC1) or placebo (normal saline) at 0, 1 and 6 months. Immediate side effects will be monitored with each visit; phone call and/or electronic check-in with daily diary for the first 8(+/-2) days post each vaccination; and blood draws to check for responses at 4 weeks post each dose and 6 months post the final dose.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The first stage will be "open-label" where 3 participants will receive the AVIHepC1 vaccine to assess for safety dosing whereas, the second stage will be double-blinded where the remaining 24 participants will receive either the AVIHepC1 vaccine or a placebo (saline).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVIHepC1 (Experimental): Contains two components: (1) GMP-Grade E1E2 heterodimer envelope protein (4.5µg); and (2) GMP-Grade SLA-SE adjuvant.
  Interventions: Biological: AVIHepC1
- Normal Saline (Placebo Comparator): 0.9% sodium chloride
  Interventions: Biological: Normal Saline

INTERVENTIONS:
Biological: AVIHepC1 — Intramuscular injection administered at 0, 4, and 24 weeks.
  Arms: AVIHepC1
Biological: Normal Saline — *Only applicable for double-blinded randomized component of the study. Intramuscular injection administered at 0, 4, and 24 weeks.
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to investigate the safety and antibody (germ fighters) response of the experimental (investigational) vaccine against HCV when injected into the arm of healthy adults.

DETAILED DESCRIPTION:
The Hepatitis C Virus (HCV) continues to be a significant public health threat, infecting 58 million people worldwide and over 250,000 Canadians. The virus disproportionately affects marginalized populations. It is a bloodborne virus that affects the liver and is most commonly spread through unsafe injection practices, sexual practices that lead to blood exposures, and unsafe health care (i.e., transfusion of contaminated blood and blood products). If left untreated, these infections progress to chronic hepatitis, liver cirrhosis (liver failure) and potentially hepatocellular carcinoma (liver cancer) or death. Current treatments for HCV include expensive drug combinations that can cure HCV in most but do not prevent reinfection if there is another exposure. At this time, there are no vaccines available to prevent HCV and the diseases that it causes.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the purpose and the procedures involved in this study and sign the informed consent form;
2. Non-pregnant individuals, 18-45 years of age inclusive;
3. Individuals must agree not to become pregnant during the trial. If they are capable of pregnancy and sexually active, they must use an effective method of birth control;
4. Non-smoker and in good general health, as determined by medical screening evaluation, performed by PI, or delegated sub-investigator no greater than 4 weeks (28 days) before the first dose in the form of medical history, clinical laboratory tests and physical examination;
5. Agrees to reside in the geographical area for next 12 months and not intending to travel outside of Canada for at least 14 days following each study vaccine administration;
6. Agree not to participate in any other clinical trial during the trial;
7. Agree not to donate blood for the duration of the trial;
8. Agree to restrain from intensive physical exercise i.e., exercise that varies significantly from an everyday exercise routine, 3 days before and after (± 3 days) administration of each dose, including each interim visit for blood sample collection;
9. Up to date on recommended seasonal vaccines (influenza and COVID-19) at the time of study enrolment.

Exclusion Criteria:

1. Presence of Hepatitis C antibody (HCV Ab);
2. Presence of significant acute infection requiring systemic antibiotic treatment within the 14 days prior to each product administration;
3. Pregnant or breast feeding (all individuals physiologically capable of pregnancy will have a negative pregnancy test result prior to each study product administered);
4. Past significant reaction following any previous vaccination;
5. History of hypersensitivity to any vaccine component;
6. Presence of acute infectious disease or fever (e.g., sub-lingual temperature 38.5°C) within the five days prior to study product administration;
7. Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immunodeficiencies), insulin dependent diabetes, progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, psoriasis, rheumatoid arthritis, asthma, epilepsy or obsessive-compulsive disorder, skin carcinoma excluding non-spreadable skin cancers such as basal cell and squamous cell carcinoma;
8. Evidence and/or any history of leukaemia, lymphoma, or neoplasm;
9. Presence or suspicion of impaired immune system function. Currently receiving or having within the past three years received immunosuppressive therapy, including systemic steroids, ACTH or inhaled steroids in dosages that are associated with hypothalamic-pituitary-adrenal axis suppression, such as 1mg/kg/day of prednisone or its equivalent or chronic use of inhaled high potency corticosteroids [budesonide 800 µg per day or fluticasone 750 µg];
10. Received blood, blood products or a parenteral immunoglobulin preparation in the past 12 weeks;
11. Evidence of bleeding diathesis or any condition that may be associated with a prolonged bleeding time;
12. Known inherited genetic anomaly (known as cytogenic disorders) e.g., Down's syndrome;
13. Evidence of any condition that, in the opinion of the clinical investigator, might interfere with the evaluation of the study objectives or pose excessive risks to participants;
14. Clinically significant abnormal laboratory as assessed by the trial physician.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 6 months after last dose of vaccine is administered
  Safety is the primary outcome. Clinical symptoms and signs, standard laboratory parameters (hematological and biochemical), and ancillary data will be collected and assessed for safety monitoring throughout the study which will also be reviewed by the Data Safety Monitoring Board (DSMB) accordingly.

SECONDARY OUTCOMES:
Immunogenicity | 6 months after last dose of vaccine is administered
  Antibody titres: Samples of sera and PBMCs will be collected from the participants prior to each injection and at the scheduled clinic visits. The titre of vaccine specific antibodies will be determined using ELISA. The presence of vaccine-specific antibodies in all participants in the study will be monitored.
Immunogenicity | 6 months after last dose of vaccine is administered
  Assessment for pan-genotypic neutralizing antibodies in vitro: Sera will be tested for neutralization capacity via a panel of infectious cell-culture-propagated HCV genotypes.
Immunogenicity | 6 months after last dose of vaccine is administered
  T cell responses: T cell responses generated by vaccinees pre- and post-vaccination will be measured by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Meier-Stephenson, MD, PhD, Study Chair — University of Alberta; Michael Houghton, PhD, Principal Investigator — University of Alberta; Lorne Tyrrell, MD, PhD, Principal Investigator — University of Alberta; Jordan Feld, MD, MSc, Principal Investigator — University of Toronto; Curtis Cooper, MD, MSc, Principal Investigator — University of Ottawa
Locations (3):
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Toronto General Hospital - Toronto Centre for Liver Disease, Toronto, Ontario